CLINICAL TRIAL: NCT03424772
Title: Clinical Collaborative Research of Whole Genome Sequencing in the Detection of Rare Undiagnosed Genetic Diseases in Children in China
Brief Title: Whole Genome Sequencing in the Detection of Rare Undiagnosed Genetic Diseases in Children in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yongguo Yu, Associate chief physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Other Study IDs: XH-18-001
Record Dates: First submitted 2018-01-30; First posted 2018-02-07 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Intellectual Disability; Multiple Congenital Anomaly; Rare Diseases
MeSH Terms: conditions — Intellectual Disability; Abnormalities, Multiple; Rare Diseases

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Genomic DNA will be extracted from whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with unexplained DD/ID: Whole genome sequencing will be performed on pediatric patients with unexplained developmental delay(DD)/intellectual disability(ID), multiple congenital abnormalities and other rare and undiagnosed diseases.
  Interventions: Diagnostic Test: Whole genome sequencing

INTERVENTIONS:
Diagnostic Test: Whole genome sequencing — WGS will be performed for the trio

SUMMARY:
To assess the indications and diagnostic efficiency of whole genome sequencing (WGS) in pediatric patients with unexplained intellectual disability/developmental delay, multiple congenital abnormalities and other rare and undiagnosed diseases

DETAILED DESCRIPTION:
This project will recruit 100 rare, undiagnosed pediatric genetic disease families (core families: patients, patients' parents, immediate family members such as brothers and sisters, all of them can be enrolled whether they have disease or not, so generally 3, for a few cases 4 or 5) all over the country. The expert team will review the clinical materials, the molecular team will review the experimental process, and the bioinformatics team will review the chip, the analysis of whole exome sequencing data and screen the samples all over the country;

Whole-genome sequencing of 100 rare, undiagnosed pediatric genetic disease families (Illumina NovaSeq High-throughput Sequencer);

The study will provide preliminarily performance data on the comparison of whole exome data and whole genome data. In addition, it will generate the Chinese Consensus on Clinical Applications of Whole-genome sequencing in the Diagnosis of Birth Defects and Undiagnosed Rare Genetic Diseases in Children based on the statistical analysis of clinical phenotype and genotype association, which could guide the clinical application of pediatrics, laboratory testing and reporting.

Construction of the Chinese detection genome database of genetic disease

ELIGIBILITY:
Inclusion Criteria:

1. Intelligence tests results of less than 40 (patients <3 years old using the Gesell Developmental Scale for screening; patients of 3-6 years old using Little Wechsler Intelligence Scale for screening; patients >6 years old using Old Wechsler Intelligence Scale for screening).
2. Neurodevelopmental defects can be expressed as mental retardation, motor development retardation, language delay, epilepsy, etc. May have or not have Multiple congenital abnormalities, families with more than one affected patient will be enrolled priority
3. Families went through at least one of the high throughput technology(WES or CMA) and receive the negative result

Exclusion Criteria:

1. Intellectual disability caused by pregnancy, perinatal infection, ischemia, and hypoxia and other non-hereditary causes,
2. Obvious genetic metabolic diseases (such as different types of genetic metabolic diseases, bone disease, fragile X syndrome, etc.);

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Undiagnosed Children with intellectual disability/developmental delay and/or multiple congenital abnormalites in China
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-01-18 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Number of diagnosed families | 1 year
  Families with rare and undiagnosed pediatric genetic disease will be benefitted by WGS.

SECONDARY OUTCOMES:
Numbers of pathogenic variants in different variation types | 1 year
  WGS would have the potential to detect different types of genetic alterations, such as structure variations, point mutation, small insertion/deletion, trinucleotide repeat, etc. Some types could not be identified by exome sequencing and chromosomal microarray. The numbers of the pathogenic variants in these types will be calculated to examine the benefit of WGS.

CONTACTS AND LOCATIONS:
Overall Officials: Yongguo Yu, MD, PhD, Principal Investigator — Specify Unaffiliated
Locations (14):
- China (14):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Children's Hospital, Capital Institute of Pediatrics, Beijing, Beijing Municipality
  - Department of Pediatrics, Peking University First Hospital, Beijing, Beijing Municipality
  - The Maternal & Child Health Hospital, The Children's Hospital, The Obstetrics & Gynecology Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Maternal and Child Health Hospital of Hunan Province, Changsha, Hunan
  - Xiangya Hospital, Central-south University / Hunan Jiahui genetics hospital, Changsha, Hunan
  - Hunan Children's Hospital, Changsha, Hunan
  - Nanjing maternal and children hospital, Nanjing, Jiangsu
  - Ruijin Hospital affiliated to Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Children's Hospital of Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Institute for Pediatric Research, Shanghai, Shanghai Municipality
  - Xin Hua Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Children's Medical Center, Shanghai, Shanghai Municipality
  - Wenzhou Central Hospital, Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
We have not yet decided which part of individual participant data(IPD) can be shared.

REFERENCES:
- [Background] Park ST, Kim J. Trends in Next-Generation Sequencing and a New Era for Whole Genome Sequencing. Int Neurourol J. 2016 Nov;20(Suppl 2):S76-83. doi: 10.5213/inj.1632742.371. Epub 2016 Nov 22. PMID 27915479
- See also: Trends in Next-Generation Sequencing and a New Era for Whole Genome Sequencing. — https://www.ncbi.nlm.nih.gov/pubmed/27915479